CLINICAL TRIAL: NCT03010982
Title: An Open-Label, Multi-Center, Two-Part, Phase 1 Study to Characterize the Pharmacokinetics of an Intravenous Micro-Dose of [14C]-Tazemetostat (EPZ 6438) and the Absorption, Distribution, Metabolism and Elimination of an Oral [14C]-Labeled Dose of Tazemetostat in Subjects With B-Cell Lymphomas or Advanced Solid Tumors
Brief Title: Open-Label, Multi-Center, Two-Part, Ph1 Study to Characterize the PKs of an Intravenous Micro-Dose of [14C]-Tazemetostat (EPZ 6438) and the ADME of an Oral [14C]-Labeled Dose of Tazemetostat in Subjects With B-Cell Lymphomas or Adv Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-103; 2016-002166-32 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2017-01-05 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Large B Cell Lymphoma; Primary Mediastinal Lymphoma; Mantle-Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Advanced Solid Tumors
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tazemetostat and [14C] Tazemetostat (Experimental): * Tazemetostat 800 mg BID orally as tablets continuously starting on Day 1, with the exception of the morning dose on Day 16;
  * A single IV dose of approximately 12 µg tazemetostat that contains approximately 500 nCi of [14C] tazemetostat on Day 15;
  * A single oral dose of 800 mg tazemetostat as a solution containing approximately 400 µCi (14.8 MBq) of [14C] tazemetostat on Day 16.
  Interventions: Drug: Tazemetostat and [14C] Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat and [14C] Tazemetostat — Tazemetostat is a selective oral small molecule inhibitor of EZH2.
  Other Names: E7438, EPZ-6438

SUMMARY:
This is a Phase 1, open-label, two-part study designed to characterize the PK of an IV dose of approximately 12 µg tazemetostat that contains approximately 500 nCi of [14C] tazemetostat and the ADME of an oral dose of 800 mg tazemetostat that contains approximately 400 µCi of [14C]-labeled tazemetostat in three subjects with B-cell lymphomas or advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age at time of consent
2. Female ≥ 18 years of age at time of consent and of non-childbearing potential. A woman is considered to be of non-childbearing potential if she has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) or has undergone surgical sterilization (removal of ovaries and/or uterus). Note: Postmenopausal state will be confirmed with FSH test completed during the screening period.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
4. Has a life expectancy of >3 months
5. Has EITHER histologically confirmed B-cell lymphomas including but not limited to diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), primary mediastinal B-cell lymphoma (PMBCL), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL), or Hodgkin lymphoma (HL) and has relapsed or refractory disease following at least two lines of prior standard therapy, including alkylator/anthracycline (unless anthracycline-based chemotherapy is contraindicated)/anti-CD20-based therapy (R-CHOP, rituximab, doxorubicin, cyclophosphamide, vincristine, and prednisolone or dexamethasone, or equivalent for non-Hodgkin lymphoma), AND must be considered unable to benefit from intensification treatment with autologous hematopoietic stem cell transplantation (ASCT) , as defined by meeting at least one of the following criteria:

   * Relapsed following, or refractory to, previous ASCT
   * Did not achieve at least a partial response to a standard salvage regimen (e.g., R-ICE, rituximab, ifosfamide, carboplatin, etoposide, or R-DHAP, rituximab, dexamethasone, cytarabine, cisplatin)
   * Ineligible for intensification treatment due to age or significant comorbidity
   * Ineligible for intensification treatment due to failure to mobilize an acceptable number of hematopoietic stem cells
   * Refused intensification treatment and/or ASCT

   OR
6. Histologically and/or cytologically confirmed advanced or metastatic solid tumor that has progressed after treatment with approved therapies or for which there are no standard therapies available
7. May have evaluable or measurable disease
8. Has all prior treatment (i.e., chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤ Grade 1 per CTCAE, version 4.03 or are clinically stable, at time of consent
9. Time between the last dose of the latest therapy and the first dose of study drug:

   1. Chemotherapy: cytotoxic - at least 21 days
   2. Chemotherapy: nitrosureas - at least 6 weeks
   3. Chemotherapy: non-cytotoxic (e.g. small molecule inhibitor) - at least 14 days
   4. Monoclonal antibody (ies) - at least 28 days
   5. Immunotherapy (e.g. tumor vaccine) - at least 28 days
   6. Radiotherapy (RT) - at least 21 days for stereotactic radiosurgery, at least 12 weeks for craniospinal, ≥50% radiation of pelvis, or total body irradiation
   7. High dose therapy with autologous hematopoietic cell infusion - at least 60 days
   8. Hematopoietic growth factor - at least 14 days
10. Has adequate hematologic (bone marrow [BM] and coagulation factors), renal and hepatic function as defined by criteria below:

    1. Hemoglobin ≥9 g/dL
    2. Platelet ≥75,000/mm3 (≥75 × 10^9/L)
    3. ANC ≥750/mm3 (≥0.75 × 10^9/L)
    4. PT< 1.5 ULN
    5. PTT< 1.5 ULN
    6. Creatinine < 2.0 ULN
    7. Conjugated bilirubin < 1.5 × ULN
    8. AST <3 × ULN I. ALT <3 × ULN NOTE: Laboratory results obtained during screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may retest the subject and the subsequent within range screening result may be used to determine the subject's eligibility
11. Subjects with a history of Hepatitis B or C are eligible on the condition that subjects have adequate liver function as defined the protocol and are hepatitis B surface antigen negative and/or have undectable HCV RNA.
12. Has a QT interval corrected by Fridericia's formula (QTcF) ≤480 msec
13. Subject must have regular bowel movements (minimum of 1 bowel movement every day or every other day; no more than 3 bowel movements per day) for the past 2 weeks without diarrhea (>4 bowel movements per day) or constipation (fewer than 3 bowel movements in 1 week). No known medical history of a disease or syndrome that affects bowel function (e.g., irritable bowel syndrome, inflammatory bowel disease, ulcerative colitis, etc.), fecal incontinence, and no history of significant opioid induced constipation within the past 3 months
14. Subject must have the ability to regularly void urine with no current evidence of urinary incontinence, urinary retention, uncorrected congenital defects that interfere with normal urinary system function, chronic urinary tract infections, or other conditions that may interfere with normal urinary bladder emptying. In the past 3 months, no obstructive uropathy, surgery affecting urinary system (e.g., radical prostatectomy, TURP, etc.), urinary tract infection. Subjects with solitary kidney are excluded from the study
15. Male subjects must refrain from donating sperm starting at the planned first dose of study drug until 30 days following the last dose of study drug. Male subjects with a female partner of childbearing potential must be vasectomized, or remain abstinent or use a condom as defined in Section 8.3.8, starting at the planned first dose of study drug until 30 days following the last dose of study drug. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Female partners of male subjects who are of childbearing potential must also adhere to one of the following:

    * Placement of an intrauterine device or intrauterine system.
    * Established use of oral, injected or implanted hormonal methods of contraception.
    * Progesterone only oral contraception, where inhibition of ovulation is not the primary mode of action.

Exclusion Criteria:

Subjects meeting ANY of the following criteria must NOT be enrolled in this study:

1. Has participated in a study in which [14C] was administered within the last 6 months prior to screening for this study
2. Has CNS or leptomeningeal metastasis
3. Has had a prior malignancy other than the malignancies under study Exception: Subject who has been disease-free for 3 years, or a subject with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible
4. Has had major surgery within 3 weeks prior to enrollment NOTE: Minor surgery (e.g., minor biopsy, central venous catheter placement) is permitted within 3 weeks prior to enrollment
5. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from time of enrollment to while on study
6. Has cardiovascular impairment, history of congestive heart failure greater than NYHA Class II uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months prior to the planned first dose of tazemetostat; or ventricular cardiac arrhythmia requiring medical treatment
7. Subjects taking medications that are known potent CYP3A4 inducers/inhibitors (including St. John's Wort) from 14 days prior to the first dose of study medications (see http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm080499.htm; or http://medicine.iupui.edu/clinpharm/ddis/ for a list of potent CYP3A4 inducers and inhibitors).
8. Has an active infection requiring systemic treatment
9. Is immunocompromised, including subjects with known history of infection with human immunodeficiency virus (HIV)
10. Has known history of chronic infection with hepatitis B virus (hepatitis B surface antigen positive) or hepatitis C virus (detectable HCV RNA)
11. Has had a venous thrombosis or pulmonary embolism within the 3 months prior to study enrollment.

    NOTE: Subjects with a history of a deep vein thrombosis >3 months prior to study enrollment who are on anticoagulation therapy with low molecular weight heparin are eligible for this study.
12. Has known hypersensitivity to any of the components of study drug
13. Is unable to take oral medications, malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea or vomiting) that might impair the bioavailability of study drug
14. Has an uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements
15. Is unwilling to adhere to contraception criteria from time of enrollment in study to at least 30 days after last dose of study drug
16. Clinical history, current alcohol (ethanol), or illicit drug use which, in the judgment of the investigator, will interfere with the subject's ability to comply with the dosing schedule and protocol-specified evaluations
17. A history of bleeding (i.e., hemoptysis, hematuria, GI blood loss, epistaxis, or others with greater than Grade 1 according to National Cancer Institute Common Terminology Criteria Version 4.0 [NCI-CTC v4.0]) within 1 month prior to beginning therapy or any clinical indications of current active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Plasma PK of [14C] tazemetostat, tazemetostat, and its metabolite EPZ-6930 after IV administration of approximately 12 µg of [14C] tazemetostat containing approximately 500 nCi of radioactivity and oral BID administration of 800 mg tazemetostat (AUC 0-7) | Day 15
Total recovery and relative excretion of radioactivity in urine and feces after an oral 800 mg dose of [14C] tazemetostat containing approximately 400 µCi (14.8 MBq) of radioactivity | Day 16

SECONDARY OUTCOMES:
Estimate tazemetostat absolute bioavailability (F) after repeated oral administration of 800 mg BID (AUC 0-12 and AUC 0-~) | Day 15
Compare the total radioactivity concentration-time profiles in blood and plasma after oral administration of [14C] tazemetostat (AUC 0-t, AUC 0-12, AUC 0-~) | Day 16
Determine peak plasma concentration (Cmax) after oral administration of [14C] tazemetostat | Day 16
Determine the plasma terminal half-life (t1/2) after oral administration of [14C] tazemetostat | Day 16
Plasma PK of tazemetostat and EPZ6930 after administration of an oral 800 mg dose of [14C] tazemetostat containing approximately 400 µCi (14.8 MBq) of radioactivity (Plasma AUC 0-t, AUC 0-12) | Day 16
Determine the peak plasma concentration (Cmax) of tazemetostat and EPZ6930 after administration of an oral 800 mg dose of [14C] tazemetostat containing approximately 400 µCi (14.8 MBq) of radioactivity | Day 16
Determine the time to peak plasma concentration (Tmax) tazemetostat and EPZ6930 after administration of an oral 800 mg dose of [14C] tazemetostat containing approximately 400 µCi (14.8 MBq) of radioactivity | Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- United Kingdom (2):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Royal Liverpool and Broadgreen University Hospital Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No